CLINICAL TRIAL: NCT00003419
Title: Treatment of HIV-Related Kaposi's Sarcoma and Stage I-III Slow-Proliferative Disease With Highly Active Antiretroviral Therapy (HAART)
Brief Title: Antiviral Therapy in Treating Patients With Slowly Progressing HIV-Related Kaposi's Sarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066438; ITA-GICAT-POS2; EU-97019
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2001-11

CONDITIONS: Sarcoma
Keywords: AIDS-related Kaposi sarcoma
MeSH Terms: conditions — Sarcoma; AIDS-related Kaposi sarcoma

INTERVENTIONS:
Procedure: antiviral therapy

SUMMARY:
RATIONALE: HIV virus is found in the lesions of most patients with Kaposi's sarcoma, and may have a role in causing Kaposi's sarcoma. Antiviral therapy acts against the HIV virus and may be an effective treatment for Kaposi's sarcoma.

PURPOSE: This phase II trial is studying how well antiviral therapy works in treating patients with slowly progressing HIV-related Kaposi's sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of highly active antiretroviral therapy (HAART) in treating patients with HIV-related stage I-III nonaggressive epidemic Kaposi's sarcoma.

OUTLINE: Patients receive therapy consisting of nucleoside analogues (RTI) and protease inhibitors (PI). Patients may receive either 2 RTIs or 2 RTIs plus 2 PIs. Treatment continues for 12 weeks, then progression is assessed.

Patients with stable or regressing Kaposi's sarcoma (KS) with a viral load of greater than 500 copies of RNA/mL may continue with the therapy (if the viral load has decreased by greater than 2 logs) or may modify therapy (if the viral load has decreased less than 2 logs). Patients with progressive disease may begin chemotherapy but continue to receive the antiretroviral therapy. Treatment continues for at least 48 weeks.

Patients are followed every 8 weeks until week 48.

PROJECTED ACCRUAL: This study will accrue a total of 14-25 patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Stage I-III (NYU) Kaposi's sarcoma that is slowly progressive

  * Stable disease without progression in diameter of tumor or in number of lesions (less than 50% increase in 3 months)
  * No progressive disease during or after treatment for Kaposi's sarcoma
* Level of viral load detectable independently from CD4+ cells
* No other active AIDS pathologies

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-3

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 1500/mm3
* Hemoglobin greater than 8 mg/dL

Hepatic:

* Bilirubin less than 2.5 times normal
* AST and ALT less than 5 times normal
* Alkaline phosphatase less than 2.5 times normal

Renal:

* Creatinine less than 2.5 times normal

Other:

* No prior malignancy except carcinoma in situ of the cervix or nonmelanomatous skin cancer
* No active cytomegalovirus, herpes simplex 1 or 2, or herpes zoster infection requiring treatment

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other

* No prior antiretroviral therapy OR
* No prior highly active antiretroviral therapy (HAART)
* No concurrent acyclovir, ganciclovir, foscarnet, or cidofovir

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 1998-06

PRIMARY OUTCOMES:
Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Tirelli, MD, Study Chair — Centro di Riferimento Oncologico - Aviano
Locations (1):
- Centro di Riferimento Oncologico - Aviano, Aviano, Italy